CLINICAL TRIAL: NCT05654246
Title: ShareForCures: Susan G. Komen's People-powered, Data-driven Breast Cancer Research Registry
Brief Title: Susan G. Komen's ShareForCures
Status: Recruiting | Type: Observational
Sponsor: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SGK-SFC-001
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — ShareForCures plans to leverage different types of biospecimens, including breast cancer tissue (retrospective), blood (retrospective and prospective), and saliva (prospective).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
ShareForCures (SFC) is a community-based participatory research registry, and its prime objective is to engage participants representative of the United States breast cancer patient population -including minoritized and historically marginalized people, persons, or communities-to ensure the data researchers use to study breast cancer is as diverse as the people touched by this disease. In doing so, researchers will have a better understanding of breast cancer, and everyone can potentially benefit from scientific advances and improvements in care.

DETAILED DESCRIPTION:
ShareForCures (SFC) will be a people-powered, data-driven breast cancer registry that will provide a way for individuals from diverse backgrounds to participate in research and enable participants' data to be used for breast cancer research. The overarching goal of SFC is to create a robust research resource comprised of clinical, biological, socio-behavioral, and other data from up to 200,000 people with breast cancer-including minoritized and historically marginalized people, persons, or communities-to ensure the data, researchers use to study breast cancer, is as diverse as the people touched by this disease. In doing so, researchers will have a better understanding of breast cancer and everyone can potentially benefit from scientific advances and improvements in care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be at least 18 years old. (Individuals in Alabama and Nebraska must be over 19 and individuals in Mississippi and Pennsylvania must be over 21 to participate).
* Individuals must have been diagnosed with cancer originating (or is suspected to originate) from the breast.
* Individuals must be currently residing in the United States or a territory of the United States.
* Individuals must be able to read and understand English.

Exclusion Criteria:

* Individuals under the age of 18 years. (Individuals in Alabama and Nebraska under 19 and individuals in Mississippi and Pennsylvania under 21 are not eligible to participate).
* Individuals without a diagnosis of breast cancer.
* Individuals who are not residing in the United States or a territory of the United States.
* Individuals unable to read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ShareForCures is open to all individuals diagnosed with breast cancer, age 18 and older, of any gender, and all racial and ethnic origins living in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Engage participants representative of the United States breast cancer patient population in ShareForCures. | 10 years
  Enroll and engage up to 200,000 people, who have been diagnosed with breast cancer, reflecting the diversity of breast cancer survivors within the United States, to participate in the registry as our partners in research.
Integrate participant data into ShareForCures. | 10 years
  Collect and curate a rich scope of participant data from a variety of sources (including participant-provided information, clinical records, and linkage to other existing datasets) and biospecimens to create a comprehensive, longitudinal database.
Facilitate scientific research using ShareForCures data. | 10 years
  Make deidentified data available to researchers for scientific discoveries, including research that may lead to new knowledge about breast cancer and advances in patient care and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Jourquin, Ph.D., M.S., Principal Investigator — Susan G. Komen
Locations (1):
- Susan G. Komen, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers may request access to SFC data, and upon approval may use the data to answer research questions including studies that will lead to new knowledge about breast cancer and advances in patient care and outcomes.
  All data sharing will be handled securely and under IRB approval or exemption, following rigorous standards to protect individual privacy and data confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: Once enough data have been aggregated in ShareForCures, researchers will be able to request access to ShareForCures deidentified data. Data will be available for the duration of the study.
Access Criteria: Researchers will be required to formally request access to the data. All requests will be reviewed according to Komen's Data Request Review Process. Researchers will also need to execute a Data Transfer and Use Agreement (DTUA), comply with the Researcher Code of Conduct, and abide by other Komen policies and procedures, as needed.
URL: https://www.komen.org/shareforcures/